CLINICAL TRIAL: NCT04078100
Title: Transseptal Approach Versus Conventional Left Atrial Approach for Mitral Valve Procedures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Beshoy Allam Moris, Dr., Assiut University
Other Study IDs: Transseptal apprroach
Record Dates: First submitted 2019-09-02; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Mitral Valve Surgical Approaches
Keywords: mitral valve replacement; transseptal approach; left atrial approach; mital valve repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: underwent mitral valve surgery through transseptal approach.
  Interventions: Procedure: Transseptal approach.
- group B: underwent mitral valve surgery through conventional left atrial approach.

INTERVENTIONS:
Procedure: Transseptal approach. — surgical approach to the mitral valve through the Fossa Ovalis by way of the right atrium.
  Groups: group A

SUMMARY:
Study Objectives/Specific Aims Overall Goal: To compare between transseptal approach and the conventional left atrial approach for mitral valve procedures.

* Objective 1: Assess the intraoperative approach related criteria in valve exposure, cardiopulmonary bypass time and intraoperative complications.
* Objective 2: Assess the outcomes and postoperative results.

DETAILED DESCRIPTION:
Mitral valve diseases are considered among the most prevalent valvular heart diseases that necessitate surgical intervention.

as the Modern international guidelines substantially recommend mitral valve repair whenever possible there is significant decrease in mitral valve replacement rates.

Cardiothoracic surgeons have to face the problem of Making a decision regarding mitral valve repair, reconstruction or replacement which requires excellent valve exposure for precise anatomical definition and manipulation taking in mind cases with specific anatomical challenges.

Since the beginning of modern cardiac surgery only two basic approaches to the mitral valve have been described by Effler who wrote in 1958 " the actual entry into the left atrium may be accomplished in either of two ways : through the Fossa Ovalis by way of the right atrium or through the posterior interatrial groove " Nowadays median sternotomy is still the most commonly used incision for mitral valve surgery which allows the best exposure for the valve through transseptal incision or through Sandergaard's groove.

Although the latter approach is the preferred method for most surgeons the transseptal approach has been revisited in more recent years in various forms by those seeking better exposure of mitral valve especially in cases with difficult anatomy.

In this paper we try to compare the transseptal approach with the conventional left atrial approach for mitral valve procedures to review previous literatures' results and to clarify the effect of using each of the two approaches in preoperative ,intra and postoperative course .

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent mitral valve replacement, mitral valve repair, redo mitral valve replacement, combined mitral and tricuspid procedures, combined mitral surgery and coronary arteries bypass graft at cardiothoracic surgery department Assiut University Hospital.

Exclusion Criteria:

* Patients with congenital mitral valve diseases .
* patient refused to sign the informed consent to be a part in the research .

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients who presented to Cardiothoracic Surgery Department, Assiut University Hospital and who meet the listed inclusion from 2016 to 2019 within the range of 100 eligible case.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
ischemic time | intraoperative registration.
  period of time from applying the aortic cross clamp till its removal in open heart surgeries during which there is no blood flow in the coronary arteries and the heart is ischemic.
whole operation time. | intraoperative registration.
  period of time from skin incision to skin closure in open heart surgery.
re-operation | with in the first 24 hrs post operative.
  re exploration through the same incision site to stop bleeding.

SECONDARY OUTCOMES:
Postoperative arrhythmias. | within the first week post operative.
  newly arising tachy or bradyarrhythmia
Hospital stay. | up to three months
  time of hospital admission postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Thabet, dr., Study Director — general surgery department, AssiutU; Mohamed Mahmoud, dr., Study Director — cardiothoracic department, AssiutU

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rezahosseini O, Rezaei M, Ahmadi Tafti SH, Jalali A, Bina P, Ghiasi A, Karimi A, Abbasi K, Shirzad M, Davoodi S, Salehi Omran A. Transseptal Approach versus Left Atrial Approach to Mitral Valve: A Propensity Score Matching Study. J Tehran Heart Cent. 2015 Oct 27;10(4):188-93. PMID 26985207
- [Background] van der Merwe J, Casselman F. Mitral Valve Replacement-Current and Future Perspectives. Open J Cardiovasc Surg. 2017 Jul 13;9:1179065217719023. doi: 10.1177/1179065217719023. eCollection 2017. PMID 28757798
- [Background] Doty JR, Caine WT. Mitral valve replacement and tricuspid valve repair through a transseptal approach for double-valve endocarditis. Multimed Man Cardiothorac Surg. 2012 Jan 1;2012:mms003. doi: 10.1093/mmcts/mms003. PMID 24414707
- [Background] Nienaber JJ, Glower DD. Minitransseptal versus left atrial approach to the mitral valve: a comparison of outcomes. Ann Thorac Surg. 2006 Sep;82(3):834-9; discussion 839. doi: 10.1016/j.athoracsur.2006.04.014. PMID 16928494
- [Background] Santibanez Escobar F, Serrano Gallardo G, Ramirez Marroquin S, Lopez Soriano F, Barragan Garcia R. The transseptal approach for mitral valve replacement revisited. Tex Heart Inst J. 1997;24(3):209-14. PMID 9339510